CLINICAL TRIAL: NCT02877823
Title: A Community-based, Family Navigator Intervention to Improve Cardiometabolic Health of Medicaid-insured Youth Identified Through an Antipsychotic Medication Preauthorization Program
Brief Title: Improving Cardiometabolic Health of Youth on Antipsychotic Medication
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Gloria Reeves, Associate Professor, Child Psychiatrist, University of Maryland, Baltimore
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 69387
Record Dates: First submitted 2016-06-07; First posted 2016-08-24 (Estimated); Last update posted 2022-10-13 (Actual); Status verified 2022-10

CONDITIONS: Childhood Obesity
Keywords: Pediatric Antipsychotic Treatment; Pediatric healthy lifestyle intervention; Parent peer support
MeSH Terms: conditions — Pediatric Obesity | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment (Experimental): 1. Home delivery of bottled water supplying 48 oz. /day for the child and 24 oz. /day per other household members (up to 6 family members).
  2. Child pedometer use and activity tracking to encourage child physical activity/goal setting and engage parents in monitoring their child's health behavior.
  3. Family Navigator Services by telephone with the parent to help engage and empower parents in child healthy lifestyle changes. They will also be able to assist with resource needs for the household (food/housing services).
  4. Healthy Lifestyle Education based on the American Academy of Pediatrics Institute for the Healthiest Childhood Weight daily guidelines which are 5 fruit and vegetable servings, two hours or less screen time, one hour or more physical activity, no sugary drinks daily and limit fruit juice to one hundred percent real fruit juice.
  Interventions: Behavioral: Treatment
- Control (Active Comparator): Healthy Lifestyle Education based on the American Academy of Pediatrics Institute for the Healthiest Childhood Weight daily guidelines which are 5 fruit and vegetable servings, two hours or less screen time, one hour or more physical activity, no sugary drinks and limit fruit juice to one hundred percent real fruit juice.
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Treatment — Healthy Lifestyle Education, bottled water, pedometer, family navigator service
  Other Names: HLE Home
  Arms: Treatment
Behavioral: Control — Healthy Lifestyle Education
  Arms: Control

SUMMARY:
Pediatric antipsychotic treatment is associated with significant obesity-related side effects, including weight gain, increased blood sugar, abnormal cholesterol, and risk of new onset diabetes. Antipsychotic-induced weight gain is most prominent over the first 6 months of treatment. In this study, youths who are started on antipsychotic medication are identified for a health intervention to minimize antipsychotic-induced weight gain and also have collateral health benefits for the child's parent. Children are identified through a Medicaid medication authorization program which provides a complete list of eligible youth. Youth-parent pairs will be enrolled. All youth and their parents enrolled in this study are offered healthy lifestyle education with simple targets to reduce risk of antipsychotic-induced weight gain (e.g. reduce sugar sweetened beverage intake, engage in 1 hour of daily physical activity). Half of families will also receive 1) home delivery of bottled water, 2) provision of a child pedometer, and 3) health coaching/support from a telephone-delivered, parent peer program (Family Navigator). Home water delivery has been demonstrated to dramatically reduce sugar sweetened beverage intake in general pediatric studies. Child pedometers will be used to encourage parent monitoring of child physical activity. Parent peer support will be provided through a Family Navigator, who is a parent with "lived experience" raising a child with special mental health needs. Family Navigators address practical barriers to lifestyle changes for low income families (e.g. identify safe environment for physical activity, support access to food pantries) and provide emotional support for parents dealing with competing child health priorities (emotional stability, obesity health concerns). Family Navigator contact is exclusively by phone, and all study visits will occur in the home. The Family Navigators are supervised by a child mental health expert team, with an on-call licensed clinician available to address any after hours/weekend urgent concerns. The impact of this intervention will be studied on both child and parent health outcomes (weight, blood pressure, sugar sweetened beverage consumption), child physical activity, as well as parent behaviors associated with child healthy lifestyle changes (e.g. modeling healthy behaviors, monitoring child activity). Assessment of the impact of this healthy lifestyle intervention on other obesity related outcomes that are monitored through blood work (e.g. blood sugar, cholesterol). These labs are obtained by community prescribers as part of standard of care and submitted to Medicaid as required for ongoing approval. No blood work will be done in this study protocol. Child lab results will be requested from the Medicaid pre-authorization program.

DETAILED DESCRIPTION:
Study Procedures:

1. Recruitment and Randomization: Eligible youths will be identified through the Maryland Peer Review program when individuals are approved for pediatric antipsychotic treatment. A complete list of all eligible youths and the head of household (parent) contact information will be provided through Medicaid. All parents will be mailed a letter to provide information on the study. The parent will be given the option to participate or opt out by phone (leave a message on a secure voicemail) or by mail (send in a response card). If parents express interest in the study or do not opt out (i.e. no response), the parent will contacted by phone to provide information and ask if they are interested in scheduling a consent visit. Consent/assent is described in consent section of this application. Intelligence quotient (IQ) screening will be completed using the Wechsler Abbreviated Scale of Intelligence and will be administered to ensure the youth has an IQ greater than 55 to determine eligibility.
2. Randomization will be performed separately in strata defined by sex and age and by sex-adjusted BMI percentile (85th percentile of BMI or below), using the permuted block method. Based on current knowledge of the population of antipsychotic treated, Medicaid-insured youths; it is anticipated that there will be more males enrolled than females.
3. Healthy Lifestyle Education (HLE) at baseline, 3 months, 6 months All participants will receive HLE, which is based on the American Academy of Pediatrics Institute for the Healthiest Childhood Weight daily guidelines which are 5 fruit/vegetable servings, 2 hours or less screen time (TV, computer time), 1 hour or more physical activity, 0 sugary drinks and limit fruit juice to 100% real fruit juice. Research staff (not a Family Navigator) will provide this teaching to all participants during home visits in order to standardize education across groups. HLE will be done at baseline, 3 months and 6 months. The parent will receive a handout with this information at each of these visits. Additionally, the research staff will demonstrate to the parent how to read food labels for beverages in the home. The parent will receive a copy of calorie count per serving for each of the beverages in the home. This step will allow us to educate families on calories of sugar sweetened beverages (SSB)and also will help us to track child access to sugar sweetened beverages in the home. Families will be given a handout that lists examples of beverages and their calorie counts per serving.
4. Study Assessments: Assessments will be completed for both the treatment and control groups as part of home visits as well as telephone calls (dietary recall) at baseline, 3 months and 6 months.

All parent/child participants:

* Weight, height, and blood pressure will be measured in the home using the same portable equipment used for our completed NIH-funded study of pharmacologic interventions for antipsychotic-induced weight gain.
* 24-hr dietary recall: Sugar sweetened beverage intake will be assessed using the United States Department of Agriculture Automated Multiple Pass Method (USDA AMPM) using National Health and Nutrition Examination Survey (NHANES) procedures. To address potential variability of SSB intake over the course of a typical week, we will follow recommended procedures to complete three 24- hour dietary recall interviews on non-consecutive days (2 weekdays, 1 weekend day) at baseline, 3 months, and 6 months. One will be completed during the home visit and the other 2 will done by telephone within one week of the study visit. Parent and child will be interviewed together to get a complete recall of the child's dietary intake over the past 24 hours.

Child-only measures

* Physical activity will be measured by accelerometry. Activity outcomes will primarily be measured with accelerometers to obtain more accurate and comprehensive assessment of activity. The same accelerometer will be secured to the child's left ankle using a hospital band for 7 day continuous measurement. The accelerometer is light weight (0.56 ounces), water proof, and small (29 mm x 37 mm). Physical activity measurements will include: 1) Estimated calorie expenditure with total accelerometer "counts"; 2) amount of time in light, moderate to vigorous, and sedentary activity. Of note, the amount of time spent in sedentary activity is an independent predictor of obesity(A pre-paid addressed Federal Express envelope will be provided to the parent to send the activity monitor back to the study team at the end of 1 week.)
* Lab results: Fasting glucose and triglyceride data will be obtained from the Maryland Peer Review Program are submitted by community providers as part of standard of care to the Maryland Peer Review Program to obtain ongoing authorization.This study protocol does not involve any phlebotomy procedures.
* Parent-only measure: 1) ENERGY-Parent Questionnaire on Parenting Practices ("ENERGY-PQ") will be used as a primary measure of parent practices/factors associated with child healthy lifestyle behaviors. The ENERGY-PQ (39) is a 121 item parent self-report measure created to assess a priori identified contributors to pediatric obesity (e.g. parent modeling). 2)Sugar sweetened beverages in the home. During home visits the parent will be asked to show any non-alcoholic beverages that are in the home so to provide teaching on reading food labels (e.g. is juice 100% fruit) and to keep track of access to sugar sweetened beverages in the home.

INTERVENTION GROUP only

1. Home delivery of bottled water: Methodology from two United States pediatric trials will be implemented by supplying 48 ounces(oz.)/day of bottled water for the child and 24 oz./day per other household members (up to 6 family members), to avoid competition for this resource and encourage healthy lifestyle practices for all family members. Bottled water will be provided for ease of storage and to encourage drinking water outside the home. All youth will be provided with a doctor's note so that they are permitted to keep a water bottle in the classroom. All families will be provided with written material that also lists benefits of tap water (fluoride for dental health, low cost), However, Baltimore City schools do not permit tap water consumption (concern about lead poisoning) and the American Academy of Pediatrics recommends bottled water as an option for parents who have concerns about quality of home water supply. The water delivery is a simple environmental intervention that is appropriate for both obese/non-obese youth.
2. Child pedometer use and activity tracking: The pedometer intervention is structured to 1) encourage child physical activity/goal setting and 2) engage parents in monitoring their child's health behavior. Youth will be given a pedometer and up to two additional replacements over the course of the study if the pedometer is lost or broken. Prior studies have raised concerns that pedometers are less accurate for overweight/obese individuals because the spring mechanism is affected by positioning (e.g. tilting at waist for individuals with large abdominal girth). However, newer design pedometers (piezo-electric internal mechanism) have improved measurements. It will be recommended to the parent that youth wear the pedometer daily and the parent will be instructed on activity monitoring and goal setting. Physical activity goals will be structured based on the "small change" approach developed by Rodearmel et al. (2007). The first two weeks the parent tracks the child's daily activity. A goal is set to increase the daily number of steps by 2000 steps over the 6-month intervention. The goal begins after the baseline steps are reviewed. The Family Navigator will assist the parent in goal setting, addressing barriers to physical activity (e.g. safe environment for play), role play how to encourage child activity, and provide emotional support to the parent in making changes. The parents will be asked to check daily child activity and record this information on a password protected, secure website (just study ID number and number of steps recorded) or call in the information on a secure voicemail and we will provide feedback on the activity at the 3- and 6- month visits (a certificate for the child with their average number of steps and a graph of mean weekly steps). Tracking steps this way rather than using a paper log will allow time stamp when the pedometer data is checked and the date and time of entries will be tracked. A secure telephone voicemail option for parents who find it difficult or cumbersome to log on to a website daily will be provided and parents receive instructions and practice of the procedure at the home visits (baseline, 3 months).
3. Family Navigator Services: Family engagement is viewed as critical to promoting youth healthy lifestyle changes. Family Navigators are viewed as "highly credible" sources of information because of their own experiences of raising a child with serious mental illness. In this study, parents will receive contact from a Family Navigator (FN) over the course of the study through both scheduled phone calls (weekly calls the first month followed by calls every 2 weeks) and ad-hoc flexible telephone delivered service (including weekend and evening call time availability). Utilization of FN services will be tracked by time, day of week, and duration of all calls. Family Navigator contact will serve to engage and empower parents in child healthy lifestyle changes. They will also be able to assist with resource needs for the household (food/housing services).

Procedures to monitor safety and minimize risks:

This study focuses on simple, behavioral targets (reduce sugar sweetened beverages, engage in daily activity) to reduce antipsychotic-induced weight gain that commonly occurs after medication treatment is initiated. Minimal risks are anticipated. A licensed child mental health clinician will be available on call (including weekends and after hours) to assess any urgent concerns reported by a participant, a Family Navigator, or a research staff member conducting a home visit. The Safety Screen will be administered with the parent and youth separately at the beginning of the visit. All staff will follow Maryland guidelines for reporting of suspected abuse/neglect, and the parents will be informed of this potential risk in confidentiality as part of the informed consent procedures. Any study charts that are needed for home visits will be transferred in a locked brief case to also protect confidentiality. Family Navigators will only have telephone contact on health coaching with a parent-guardian. Other adult family members who have a caregiver role (e.g. grandparent) can participate in a call only if invited by the parent and only when the parent is on the call (e.g. a parent can opt to include someone else by speaker phone). If the parent requests to have another caregiver join the visit or call no assessments or procedures will be conducted with that person and they will not be consented. The only purpose for allowing them to join a call or visit is to support the parent/child participants. Prior to signing consent, the Confirmation of Participant Understanding of Consent form will be administered. If the parent does not verbalize an adequate understanding of the study the research assistant (RA) will review the consent again with the parent, answer questions and then re-administer the Confirmation of Participant Understanding of Consent Form. If the parent is still unable to verbalize an adequate understanding of the study the Principal Investigator will meet with the parent to determine if they have an adequate understanding to be eligible to participate. If the parent does not verbalize an adequate understanding of the study they will not be eligible to participate.

The Safety monitor will be notified within 48 hours of 1) any adverse events, including patient use of emergency services (Emergency room visits, hospitalizations) 2) any Child Protective Services reports; or 3) any clinically urgent concerns assessed by the on-call clinician (e.g. clinician called because parent's blood pressure met flag for review by a medical provider on our team).

ELIGIBILITY:
Inclusion Criteria:

1. Youth between the ages of 8-16 (inclusive) at time of enrollment
2. New antipsychotic prescription preauthorization approval in the Maryland Medicaid Peer Review program (youth)
3. Parent/legal guardian of the eligible youth

Exclusion Criteria:

1. One or both of dyad pair is non-English speaking
2. Youth lacking parent/ guardian with authority to consent for treatment (foster care youth)
3. Youth residing in residential, group home, or juvenile justice detention facilities (parent participation is required to support daily activity goals)
4. Youth currently treated in an inpatient hospital treatment program
5. Youth unable to communicate verbally (to participate in dietary recall)
6. Youth IQ <55 by WASI
7. Youth who are wheelchair bound (due to accelerometer placement)

Ages: 8 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 302 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Change in youth BMI z-score from baseline to 6 months | baseline, 3 months, 6 months
  Measurement of height/weight to calculate BMI and conversion to z-score at baseline, 3 months, 6 month
Change in youth sugar sweetened beverage consumption | baseline, 3 months, 6 months
  USDA 24 hour dietary recall administered at baseline, 3 months and 6 months
Change in youth physical activity level | baseline, 3 months, 6 months
  Measured by accelerometry for 1 week at baseline, 3 months, 6 months

SECONDARY OUTCOMES:
Change in parent BMI | baseline, 3 months,6 months
  Measurement of height/weight at baseline, 3 months, 6 months
Change in parent activity level | baseline, 3 months,6 months
  Measured by the ENERGY-Parent Questionnaire at baseline, 3 month, 6 month
Change in parent consumption of sugar sweetened beverages (SSB) | baseline, 3 months, 6 months
  USDA 24 hour dietary recall at baseline, 3 months, 6 months
Change in parent blood pressure (BP) | baseline, 3 months, 6 months
  BP at baseline, 3 months, 6 months

OTHER OUTCOMES:
Change in youth blood pressure | baseline, 3 months,6 months
  Measure blood pressure at baseline, 3 and 6 months.
Change in youth fasting glucose from baseline to 6 months | baseline, 3 months,6 months
  fasting glucose at baseline, 3 months, 6 months
Change in youth fasting triglycerides from baseline to 6 months | baseline, 3 months, 6 months
  fasting triglycerides at baseline, 3 months, 6 months

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Christian RB, Gaynes BN, Saavedra LM, Sheitman B, Wines R, Jonas DE, Viswanathan M, Ellis AR, Woodell C, Carey TS. Use of antipsychotic medications in pediatric and young adult populations: future research needs. J Psychiatr Pract. 2015 Jan;21(1):26-36. doi: 10.1097/01.pra.0000460619.10429.4c. PMID 25603449
- [Result] Ogden CL, Carroll MD, Kit BK, Flegal KM. Prevalence of childhood and adult obesity in the United States, 2011-2012. JAMA. 2014 Feb 26;311(8):806-14. doi: 10.1001/jama.2014.732. PMID 24570244
- [Result] Juonala M, Magnussen CG, Berenson GS, Venn A, Burns TL, Sabin MA, Srinivasan SR, Daniels SR, Davis PH, Chen W, Sun C, Cheung M, Viikari JS, Dwyer T, Raitakari OT. Childhood adiposity, adult adiposity, and cardiovascular risk factors. N Engl J Med. 2011 Nov 17;365(20):1876-85. doi: 10.1056/NEJMoa1010112. PMID 22087679
- [Result] Olfson M, Blanco C, Liu SM, Wang S, Correll CU. National trends in the office-based treatment of children, adolescents, and adults with antipsychotics. Arch Gen Psychiatry. 2012 Dec;69(12):1247-56. doi: 10.1001/archgenpsychiatry.2012.647. PMID 22868273
- [Result] Skinner AC, Steiner MJ, Perrin EM. Self-reported energy intake by age in overweight and healthy-weight children in NHANES, 2001-2008. Pediatrics. 2012 Oct;130(4):e936-42. doi: 10.1542/peds.2012-0605. Epub 2012 Sep 10. PMID 22966024
- [Result] Borrud L, Chiappa MM, Burt VL, Gahche J, Zipf G, Johnson CL, Dohrmann SM. National Health and Nutrition Examination Survey: national youth fitness survey plan, operations, and analysis, 2012. Vital Health Stat 2. 2014 Apr;(163):1-24. PMID 24709592
- [Result] Correll CU, Manu P, Olshanskiy V, Napolitano B, Kane JM, Malhotra AK. Cardiometabolic risk of second-generation antipsychotic medications during first-time use in children and adolescents. JAMA. 2009 Oct 28;302(16):1765-73. doi: 10.1001/jama.2009.1549. PMID 19861668
- [Result] Bushe CJ, Slooff CJ, Haddad PM, Karagianis JL. Weight change from 3-year observational data: findings from the worldwide schizophrenia outpatient health outcomes database. J Clin Psychiatry. 2012 Jun;73(6):e749-55. doi: 10.4088/JCP.11m07246. PMID 22795214
- [Result] Ballon JS, Pajvani U, Freyberg Z, Leibel RL, Lieberman JA. Molecular pathophysiology of metabolic effects of antipsychotic medications. Trends Endocrinol Metab. 2014 Nov;25(11):593-600. doi: 10.1016/j.tem.2014.07.004. Epub 2014 Sep 2. PMID 25190097
- [Result] Cote AT, Devlin AM, Panagiotopoulos C. Initial screening of children treated with second-generation antipsychotics points to an association between physical activity and insulin resistance. Pediatr Exerc Sci. 2014 Nov;26(4):455-62. doi: 10.1123/pes.2014-0076. PMID 25372380
- [Result] De Hert M, Dobbelaere M, Sheridan EM, Cohen D, Correll CU. Metabolic and endocrine adverse effects of second-generation antipsychotics in children and adolescents: A systematic review of randomized, placebo controlled trials and guidelines for clinical practice. Eur Psychiatry. 2011 Apr;26(3):144-58. doi: 10.1016/j.eurpsy.2010.09.011. Epub 2011 Feb 3. PMID 21295450
- [Result] Lipscombe LL, Austin PC, Alessi-Severini S, Blackburn DF, Blais L, Bresee L, Filion KB, Kawasumi Y, Kurdyak P, Platt RW, Tamim H, Paterson JM; Canadian Network for Observational Drug Effect Studies (CNODES) Investigators. Atypical antipsychotics and hyperglycemic emergencies: multicentre, retrospective cohort study of administrative data. Schizophr Res. 2014 Apr;154(1-3):54-60. doi: 10.1016/j.schres.2014.01.043. Epub 2014 Feb 24. PMID 24581419
- [Result] Delpier T, Giordana S, Wedin BM. Decreasing sugar-sweetened beverage consumption in the rural adolescent population. J Pediatr Health Care. 2013 Nov-Dec;27(6):470-8. doi: 10.1016/j.pedhc.2012.07.002. Epub 2012 Aug 26. PMID 22932228
- [Result] Miller PE, McKinnon RA, Krebs-Smith SM, Subar AF, Chriqui J, Kahle L, Reedy J. Sugar-sweetened beverage consumption in the U.S.: novel assessment methodology. Am J Prev Med. 2013 Oct;45(4):416-21. doi: 10.1016/j.amepre.2013.05.014. PMID 24050417
- [Result] Basu S, Seligman HK, Gardner C, Bhattacharya J. Ending SNAP subsidies for sugar-sweetened beverages could reduce obesity and type 2 diabetes. Health Aff (Millwood). 2014 Jun;33(6):1032-9. doi: 10.1377/hlthaff.2013.1246. PMID 24889953
- [Result] Wang YC, Bleich SN, Gortmaker SL. Increasing caloric contribution from sugar-sweetened beverages and 100% fruit juices among US children and adolescents, 1988-2004. Pediatrics. 2008 Jun;121(6):e1604-14. doi: 10.1542/peds.2007-2834. PMID 18519465
- [Result] Johnson RK, Appel LJ, Brands M, Howard BV, Lefevre M, Lustig RH, Sacks F, Steffen LM, Wylie-Rosett J; American Heart Association Nutrition Committee of the Council on Nutrition, Physical Activity, and Metabolism and the Council on Epidemiology and Prevention. Dietary sugars intake and cardiovascular health: a scientific statement from the American Heart Association. Circulation. 2009 Sep 15;120(11):1011-20. doi: 10.1161/CIRCULATIONAHA.109.192627. Epub 2009 Aug 24. PMID 19704096
- [Result] Stanhope KL, Medici V, Bremer AA, Lee V, Lam HD, Nunez MV, Chen GX, Keim NL, Havel PJ. A dose-response study of consuming high-fructose corn syrup-sweetened beverages on lipid/lipoprotein risk factors for cardiovascular disease in young adults. Am J Clin Nutr. 2015 Jun;101(6):1144-54. doi: 10.3945/ajcn.114.100461. Epub 2015 Apr 22. PMID 25904601
- [Result] Ebbeling CB, Feldman HA, Osganian SK, Chomitz VR, Ellenbogen SJ, Ludwig DS. Effects of decreasing sugar-sweetened beverage consumption on body weight in adolescents: a randomized, controlled pilot study. Pediatrics. 2006 Mar;117(3):673-80. doi: 10.1542/peds.2005-0983. PMID 16510646
- [Result] Ebbeling CB, Feldman HA, Chomitz VR, Antonelli TA, Gortmaker SL, Osganian SK, Ludwig DS. A randomized trial of sugar-sweetened beverages and adolescent body weight. N Engl J Med. 2012 Oct 11;367(15):1407-16. doi: 10.1056/NEJMoa1203388. Epub 2012 Sep 21. PMID 22998339
- [Result] Tate DF, Turner-McGrievy G, Lyons E, Stevens J, Erickson K, Polzien K, Diamond M, Wang X, Popkin B. Replacing caloric beverages with water or diet beverages for weight loss in adults: main results of the Choose Healthy Options Consciously Everyday (CHOICE) randomized clinical trial. Am J Clin Nutr. 2012 Mar;95(3):555-63. doi: 10.3945/ajcn.111.026278. Epub 2012 Feb 1. PMID 22301929
- [Result] Ho M, Garnett SP, Baur LA, Burrows T, Stewart L, Neve M, Collins C. Impact of dietary and exercise interventions on weight change and metabolic outcomes in obese children and adolescents: a systematic review and meta-analysis of randomized trials. JAMA Pediatr. 2013 Aug 1;167(8):759-68. doi: 10.1001/jamapediatrics.2013.1453. PMID 23778747
- [Result] Tandon PS, Zhou C, Sallis JF, Cain KL, Frank LD, Saelens BE. Home environment relationships with children's physical activity, sedentary time, and screen time by socioeconomic status. Int J Behav Nutr Phys Act. 2012 Jul 26;9:88. doi: 10.1186/1479-5868-9-88. PMID 22835155
- [Result] Rodearmel SJ, Wyatt HR, Stroebele N, Smith SM, Ogden LG, Hill JO. Small changes in dietary sugar and physical activity as an approach to preventing excessive weight gain: the America on the Move family study. Pediatrics. 2007 Oct;120(4):e869-79. doi: 10.1542/peds.2006-2927. PMID 17908743
- [Result] Janicke DM, Steele RG, Gayes LA, Lim CS, Clifford LM, Schneider EM, Carmody JK, Westen S. Systematic review and meta-analysis of comprehensive behavioral family lifestyle interventions addressing pediatric obesity. J Pediatr Psychol. 2014 Sep;39(8):809-25. doi: 10.1093/jpepsy/jsu023. Epub 2014 May 13. PMID 24824614
- [Result] Van Lippevelde W, te Velde SJ, Verloigne M, De Bourdeaudhuij I, Manios Y, Bere E, Jan N, Fernandez-Alvira JM, Chinapaw MJ, Bringolf-Isler B, Kovacs E, Brug J, Maes L. Associations between home- and family-related factors and fruit juice and soft drink intake among 10- to 12-year old children. The ENERGY project. Appetite. 2013 Feb;61(1):59-65. doi: 10.1016/j.appet.2012.10.019. Epub 2012 Nov 12. PMID 23154218
- [Result] Skelton JA, Buehler C, Irby MB, Grzywacz JG. Where are family theories in family-based obesity treatment?: conceptualizing the study of families in pediatric weight management. Int J Obes (Lond). 2012 Jul;36(7):891-900. doi: 10.1038/ijo.2012.56. Epub 2012 Apr 24. PMID 22531090
- [Result] Reeves GM, Keeton C, Correll CU, Johnson JL, Hamer RM, Sikich L, Hazzard L, Alderman C, Scheer A, Mabe M, Kapoor S, Sheridan E, Borner I, Bussell K, Pirmohamed S, Bethea TC, Chekuri R, Gottfried R, Reinblatt SP, Santana E, Riddle MA. Improving metabolic parameters of antipsychotic child treatment (IMPACT) study: rationale, design, and methods. Child Adolesc Psychiatry Ment Health. 2013 Aug 15;7(1):31. doi: 10.1186/1753-2000-7-31. PMID 23947389
- [Result] Gohlke JM, Dhurandhar EJ, Correll CU, Morrato EH, Newcomer JW, Remington G, Nasrallah HA, Crystal S, Nicol G; Adipogenic and Metabolic Effects of APDs Conference Speakers; Allison DB. Recent advances in understanding and mitigating adipogenic and metabolic effects of antipsychotic drugs. Front Psychiatry. 2012 Jun 28;3:62. doi: 10.3389/fpsyt.2012.00062. eCollection 2012. PMID 22754543
- [Result] Trapp GS, Giles-Corti B, Bulsara M, Christian HE, Timperio AF, McCormack GR, Villanueva K. Measurement of children's physical activity using a pedometer with a built-in memory. J Sci Med Sport. 2013 May;16(3):222-6. doi: 10.1016/j.jsams.2012.06.011. Epub 2012 Jul 31. PMID 22854294
- [Result] Singh AS, Chinapaw MJ, Uijtdewilligen L, Vik FN, van Lippevelde W, Fernandez-Alvira JM, Stomfai S, Manios Y, van der Sluijs M, Terwee C, Brug J. Test-retest reliability and construct validity of the ENERGY-parent questionnaire on parenting practices, energy balance-related behaviours and their potential behavioural determinants: the ENERGY-project. BMC Res Notes. 2012 Aug 13;5:434. doi: 10.1186/1756-0500-5-434. PMID 22888983
- [Result] Reeves GM, Wehring HJ, Connors KM, Bussell K, Schiffman J, Medoff DR, Tsuji T, Walker J, Brown A, Strobeck D, Clough T, Rush CB, Riddle MA, Love RC, Zachik A, Hoagwood K, Olin SS, Stephan S, Okuzawa N, Edwards S, Baquet C, dosReis S. The Family Value of Information, Community Support, and Experience Study: Rationale, Design, and Methods of a "Family-Centered" Research Study. J Nerv Ment Dis. 2015 Dec;203(12):896-900. doi: 10.1097/NMD.0000000000000393. PMID 26524515
- [Derived] Bussell K, Reeves G, Hager E, Zhu S, Correll CU, Riddle MA, Sikich L. Dietary Consumption Among Youth with Antipsychotic-Induced Weight Gain and Changes Following Healthy Lifestyle Education. J Child Adolesc Psychopharmacol. 2021 Jun;31(5):364-375. doi: 10.1089/cap.2020.0173. PMID 34143682